CLINICAL TRIAL: NCT02550678
Title: A Phase 1/2a Study of the Efficacy and Safety of ASN-002 Alone or in Combination With 5-FU in Adult Patients With Low-risk Nodular Basal Cell Carcinoma
Brief Title: A Study of the Efficacy and Safety of ASN-002 in Adult Patients With Low-risk Nodular Basal Cell Carcinoma
Acronym: ASN-002-001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascend Biopharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASN-002-001
Record Dates: First submitted 2015-09-10; First posted 2015-09-15 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Basal Cell Nevus Syndrome; Skin Neoplasm; Nodular Basal Cell Carcinoma of Skin
Keywords: Untreated nBCC; Low-Risk
MeSH Terms: conditions — Basal Cell Nevus Syndrome; Skin Neoplasms | interventions — gusacitinib; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Study Participants will receive ASN-002 at a dose 5X 10(10) vp, weekly injection in tumor nodules for 3 weeks.
  Interventions: Biological: ASN-002
- Cohort 2 (Experimental): Study Participants will receive ASN-002 at a dose of 1.5X 10(11) vp weekly injection in tumor nodules for 3 weeks
  Interventions: Biological: ASN-002
- Cohort 4 (Experimental): Study Participants will receive ASN- 002 at a dose of 3.0X 10(11) vp weekly injections in tumor nodules for 3 weeks.
  Interventions: Biological: ASN-002
- Cohort 5 (Experimental): Study Participants will receive ASN- 002 at a dose of 2.25X 10(11) vp weekly injections in tumor nodules for 3 weeks.
  Interventions: Biological: ASN-002
- Combination Cohorts (Experimental): Study Participants will receive ASN- 002 at either dose of Cohorts II, IV or V in combination with a low dose 5-FU (1mg/2.5 mg/5mg/10mg or 25mg) weekly injections in tumor nodules for 3 weeks.
  Interventions: Biological: ASN-002; Drug: 5-FU

INTERVENTIONS:
Biological: ASN-002 — ASN-002, is made of a suspension of recombinant adenoviral particles carrying a gene coding for the human interferon-gamma (IFN). Study participants will receive protocol defined dose of ASN-002 as intra-tumoral injections.
Drug: 5-FU — 5-FU is chemotherapeutic agent used to treat various cancers.
  Arms: Combination Cohorts

SUMMARY:
The study evaluates whether ASN-002 is safe and effective in the treatment of nodular basal cell carcinoma (nBCC) in patients aged 18 years or over.

The participants will receive weekly injections of ASN-002 alone or in combination with 5-FU for 3 weeks and undergo surgical excision of the tumor.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine whether ASN-002 alone or in combination with 5-FU is safe and effective in the treatment of nodular basal cell carcinoma (nBCC).

Patients aged 18 or over, who have been diagnosed with nodular Basal Cell Carcinoma (nBCC), may be eligible to join this study.

Study details:

ASN-002 is an immunotherapeutic product that is injected into the BCC spot to be treated. It is made from modified adenovirus serotype 5 (also called Ad5). Adenoviruses are common in nature worldwide and can cause mild colds and respiratory infections from which people usually recover without treatment. The Ad5 used in this study has been modified so that it cannot grow in the body or cause an infection. The modified Ad5 in this study will deliver artificially made genetic material into the cancerous and surrounding cells. This genetic material will produce human interferon which is normally produced by the body to stimulate the immune system. It is hoped that injected ASN-002 will cause the body's own cells to produce interferon and stimulate the immune system to attack the cancerous cells and reduce the size of or eliminate the nBCC. Participants will attend the study centre weekly for an injection of ASN-002 alone of in combination with 5-FU into the nBCC. The participants recruited will have 3 injections over 3 weeks, and then undergo surgical excision of the tumor.

Patient outcomes will then be assessed using a tumour sample collected during surgery and by the incidence of adverse events which occur throughout the study.

It is hoped that the findings of this trial will provide information on the safety and efficacy of using ASN-002 alone or in combination with 5-FU for nBCC, particularly for patients in whom the standard treatment of surgery is not possible or not recommended.

ELIGIBILITY:
Inclusion Criteria:

1. Low risk nodular basal cell carcinoma
2. Biopsy of any other skin tumor
3. Willingness to have injection therapy followed by surgery
4. Written informed consent

Exclusion Criteria:

1. No or only minimal symptoms
2. Known or suspected metastatic disease.
3. Pregnant or Lactating females
4. Clinically active or uncontrolled skin disease
5. Immunocompromised or receiving immunomodulating agent
6. treatment with psoralen plus Ultraviolet A or Ultraviolet B light therapy within 6 months
7. Any serious or active medical or psychiatric illness
8. Recreational or therapeutic drug or alcohol use
9. Taking any investigational product within 1 month of first dose of ASN- 002.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Incidences of ASN-002 related Adverse Event in patients with previously untreated nBCC | Participants will be followed up for up to 6 months.
  changes in vital signs, adverse events, serious adverse events, laboratory abnormalities and withdrawals from study. Local skin and injection site reactions will be assessed in detail scoring erythema, ulceration, pain and overall severity as none, mild, moderate or severe.

SECONDARY OUTCOMES:
Microscopic clearance of the injected basal cell carcinoma. | Microscopic examinations of sample collected at 17weeks after the first dose.
  Histological clearance (HC) will be defined as the absence of detectable evidence of BCC tumor cell nests in serial histological samples as determined by central pathology review.
Clinical Changes in size of nBCC tumor over time after treatment with ASN-002 alone or in combination with 5-FU | Change in nBCC will be assessed for up to 6 months from the first treatment visit.
  Change in nBCC lesion size will be assessed by investigator at baseline and then every 4 weeks until the surgical excision of BCC after ASN-002 therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Spelman, Principal Investigator — Veracity Clinical Research Pty Ltd.; Rodney Sinclair, Principal Investigator — Sinclair Dermatology Pty Ltd; Gregory Siller, Principal Investigator — Siller Medical T/A Central Brisbane Dermatology
Locations (4):
- Australia (4):
  - St George Dermatology and Skin Cancer Centre, Kogarah, New South Wales
  - Siller Medical T/A Central Brisbane Dermatology, Brisbane, Queensland
  - Veracity Clinical Research, Brisbane, Queensland
  - Sinclair Dermatology, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No